CLINICAL TRIAL: NCT00102973
Title: Phase III Randomized Study of TLK286 (Telcyta) in Combination With Carboplatin (Paraplatin) Versus Liposomal Doxorubicin (Doxil) as Second-Line Therapy in Platinum Refractory or Resistant Ovarian Cancer [ASSIST-3]
Brief Title: TLK286 (Telcyta) in Combination With Carboplatin (Paraplatin) Versus Doxil in Platinum Refractory or Resistant Ovarian Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Telik (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TLK286.3024
Record Dates: First submitted 2005-02-04; First posted 2005-02-07 (Estimated); Last update posted 2012-05-31 (Estimated); Status verified 2006-06

CONDITIONS: Ovarian Neoplasms
Keywords: Ovary
MeSH Terms: conditions — Ovarian Neoplasms | interventions — TER 286; Carboplatin

ARMS (2):
- TLK286 in Combination with Carboplatin (Experimental)
  Interventions: Drug: TLK286 in Combination with Carboplatin
- Doxorubisin HCl Liposome Injection (Active Comparator)
  Interventions: Drug: Doxorubicin HCl Liposome Injection

INTERVENTIONS:
Drug: TLK286 in Combination with Carboplatin — Experimental Arm
  Arms: TLK286 in Combination with Carboplatin
Drug: Doxorubicin HCl Liposome Injection — Active Comparator
  Arms: Doxorubisin HCl Liposome Injection

SUMMARY:
The purpose of this research study is to determine if TLK286 given in combination with carboplatin is more effective than liposomal doxorubicin in treating women who have recurrent ovarian epithelial cancer, fallopian tube cancer, or primary peritoneal cancer, that is refractory or resistant to platinum chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Are a woman 18 years of age or older
* Have histologically or cytologically confirmed epithelial cancer of the ovary or fallopian tube, or primary peritoneal cancer
* Have platinum refractory or resistant cancer
* Measurable disease according to radiographic RECIST criteria with documented tumor progression

Exclusion Criteria:

* Had treatment with first-line chemotherapy other than platinum-based regimens (carboplatin or cisplatin)
* Have clinically significant cardiac disease
* Have any sign of intestinal obstruction interfering with nutrition at the time of study entry
* Are pregnant or lactating
* Had prior treatment with liposomal doxorubicin for ovarian cancer
* Had prior treatment with TLK286

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2004-12; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Study Objectives | Every 8 Weeks
  To demonstrate superiority in the objective response rate (ORR) of TLK286 in combination with carboplatin as compared to active control therapy with liposomal doxorubicin

CONTACTS AND LOCATIONS:
Locations (216):
- United States (216):
  - Little Rock Hematology Oncology, Little Rock, Arkansas
  - Arkansas Oncology Associates, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Anaheim, California
  - East Bay Oncology/Hematology Medical Associates, Inc., Antioch, California
  - Southern California Permanente Medical Group, Baldwin Park, California
  - Southern California Permanente Medical Group, Bellflower, California
  - Marilyn Norton, M.D., Chula Vista, California
  - Bay Area Cancer Research Group, LLC, Concord, California
  - East Bay Oncology/Hematology Medical Associates, Inc., Concord, California
  - Southwest Cancer Care, Escondido, California
  - Southern California Permanente Medical Group, Fontana, California
  - California Oncology of the Central Valley, Fresno, California
  - Southern California Permanente Medical Group, Harbor City, California
  - Kaiser Permanente Medical Center, Hayward, California
  - Gynecologic Oncology Associates, La Jolla, California
  - Cancer Center Oncology Medical Group, La Mesa, California
  - LLU Faculty Medical Offices, Loma Linda, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Southern California Permanente Medical Group, Los Angeles, California
  - Bowyer Oncology Center, Los Angeles, California
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - OB/GYN Consult Suite, Los Angeles, California
  - Beverly Oncology and Imaging, Montebello, California
  - Clinical Trials and Research Associates, Inc., Montebello, California
  - Oncology Care Medical Associates, Montebello, California
  - Southwest Cancer Care, Murrieta, California
  - Newport Imaging Center, Newport Beach, California
  - Gynecologic Oncology Associates, Newport Beach, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Kaiser Permanente Medical Center, Oakland, California
  - N. County Oncology Medical, Oceanside, California
  - Southern California Permanente Medical Group, Panorama City, California
  - Southwest Cancer Care, Poway, California
  - Southern California Permanente Medical Group, Riverside, California
  - Kaiser Permanente Medical Center, Sacramento, California
  - Medical Oncology Associates, San Diego, California
  - Sharp Memorial Hospital - Investigational Pharmacy, San Diego, California
  - Sharp Rees-Stealy, San Diego, California
  - Kaiser Permanente Medical Center, San Francisco, California
  - Oncology Care Medical Associates, San Gabriel, California
  - Kaiser Permanente Medical Center, San Jose, California
  - Kaiser Permanente Medical Center, Santa Clara, California
  - Kaiser Permanente Medical Center, South San Francisco, California
  - Kaiser Permanente Medical Center, Vallejo, California
  - Kaiser Permanente Medical Center, Walnut Creek, California
  - Diablo Valley Oncology & Hematology Medical Group, Inc., Walnut Creek, California
  - Oncology Care Medical Associates, Whittier, California
  - Southern Permanente Medical Group, Woodland Hills, California
  - University of Connecticut Health Center/John Dempsey Hospital, Farmington, Connecticut
  - The Center for Hematology-Oncology, Boca Raton, Florida
  - Citrus Diagnostic Center, Crystal River, Florida
  - Citrus Hematology and Oncology Center, Crystal River, Florida
  - The Center for Hematology-Oncology, Delray Beach, Florida
  - GYN Oncology Associates, Inc., Hollywood, Florida
  - Citrus Hematology and Oncology Center, Inverness, Florida
  - Citrus Memorial Hospital Radiology Dept., Inverness, Florida
  - Florida Wellcare Alliance, LC, Inverness, Florida
  - Shands Jacksonville Medical Center, Jacksonville, Florida
  - Palm Beach Cancer Institute, Jupiter, Florida
  - Cancer and Blood Disease Center, Lecanto, Florida
  - Florida Hospital, Orlando, Florida
  - Gynecology Oncology, Orlando, Florida
  - Florida Hospital Memorial Division - Cancer Care Center, Ormond Beach, Florida
  - Florida Hospital Memorial System, Ormond Beach, Florida
  - Palm Beach Cancer Institute, Palm Beach Gardens, Florida
  - GYN Oncology Associates, Inc., Pembroke Pines, Florida
  - Palm Beach Cancer Institute, Wellington, Florida
  - Palm Beach Cancer Institute, West Palm Beach, Florida
  - Southeastern Gynecologic Oncology, Atlanta, Georgia
  - Southeastern Gynecologic Oncology, Lawrenceville, Georgia
  - Southeastern Gynecologic Oncology, Marietta, Georgia
  - Southeastern Gynecologic Oncology, Riverdale, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Southeastern Gynecologic Oncology, Tucker, Georgia
  - Kaiser Permanente Hawaii, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Joliet Oncology-Hematology Associates, Inc., Flossmoor, Illinois
  - Joliet Oncology-Hematology Associates, Inc., Joliet, Illinois
  - Joliet Oncology-Hematology Associates, Inc., Kankakee, Illinois
  - Joliet Oncology-Hematology Associates, Inc., Morris, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - St. Vincent Hospital, Indianapolis, Indiana
  - LaPorte Hospital, La Porte, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph's Regional Medical Center, South Bend, Indiana
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - University Medical Center, Inc. DBA: U of L Hospital, Louisville, Kentucky
  - Hematology and Oncology Specialists, LLC, Covington, Louisiana
  - OncRx (Pharmacy), Metairie, Louisiana
  - Hematology and Oncology Specialist, New Orleans, Louisiana
  - LSU Health Sciences Center, Shreveport, Louisiana
  - Maine Medical Center - Brighton Campus, Portland, Maine
  - Maine Medical Center, Portland, Maine
  - Maine Medical Center - Scarborough Campus, Scarborough, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Center for Cancer and Blood Disorders, P. C., Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber/Partners Cancer Care, Inc., Boston, Massachusetts
  - Boston Medical Center - Center for Cancer and Blood Disorders, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Caritas St. Elizabeth's Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Perceptive Informatics, Inc., Waltham, Massachusetts
  - Sparrow Health System, Lansing, Michigan
  - Lakeland Hospital, Niles, Michigan
  - Lakeland Hospital, Saint Joseph, Michigan
  - Providence Cancer Institute and Hospital, Southfield, Michigan
  - Duluth Clinic, Duluth, Minnesota
  - The Family Cancer Center, Olive Branch, Mississippi
  - Ellis Fischel Cancer Center, Columbia, Missouri
  - Saint Louis University, St Louis, Missouri
  - St. John's Mercy Medical Center, St Louis, Missouri
  - St. John's Mercy-David C. Pratt Cancer Center, St Louis, Missouri
  - Deaconess Billings Clinic, Billings, Montana
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology & Oncology Consultants, PC, Omaha, Nebraska
  - Horizons West Medical Group, Scottsbluff, Nebraska
  - Odyssey Research, Scottsbluff, Nebraska
  - Regional West Medical Center, Scottsbluff, Nebraska
  - The Women's Center of Western Nebraska, Scottsbluff, Nebraska
  - Mary Hitchcock Memorial Hospital/Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - A. Richard Miskoff, DO, PA, Edison, New Jersey
  - JFK Medical Center, Edison, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - The Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Jsumc Ob/Gyn, West Long Branch, New Jersey
  - Gynecologic Oncology & Minimally Invasive Surgery, Babylon, New York
  - The Mary Imogene Bassett Hospital, Cooperstown, New York
  - Schwartz Gynecologic Oncology, East Islip, New York
  - North Shore University Hospital, Manhasset, New York
  - Hematology-Oncology Associates of Rockland, New City, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - The Union State Bank Cancer Center, Nyack, New York
  - Asheville Radiology, Asheville, North Carolina
  - Hope A Women's Cancer Center, Asheville, North Carolina
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Inpatient Pharmacy, Charlotte, North Carolina
  - Blumenthal Cancer Center, Charlotte, North Carolina
  - Presbyterian Gynecologic Oncology, Charlotte, North Carolina
  - Presbyterian Hospital, Charlotte, North Carolina
  - Piedmont Hematology Oncology Associates, Winston-Salem, North Carolina
  - Cancer Care Center - Medcenter One, Inc., Bismarck, North Dakota
  - Cancer Treatment & Research Center - Mid Dakota Clinic, P. C., Bismarck, North Dakota
  - Odyssey Research, Bismarck, North Dakota
  - Dakota Cancer Institute, Fargo, North Dakota
  - Odyssey Research, Fargo, North Dakota
  - Barrett Cancer Center, Cincinnati, Ohio
  - UC Physician's Medical Arts Building, Cincinnati, Ohio
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Fairview Hospital Moll Pavilion, Cleveland, Ohio
  - Mid Ohio Onc/Hem (East), Columbus, Ohio
  - GOPSA, Columbus, Ohio
  - Mid Ohio Onc/Hem (West), Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Hillcrest Hospital/Cleveland Clinic Health System, Mayfield Heights, Ohio
  - Garth Phibbs, M.D., FACOG, Toledo, Ohio
  - ProMedica Health System, Toledo, Ohio
  - The Toledo Hospital, Toledo, Ohio
  - Mid Onio Onc/Hem (North), Westerville, Ohio
  - Cancer Care Associates, Tulsa, Oklahoma
  - Kaiser Permanente Northwest Region, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Advance Imaging, Dunmore, Pennsylvania
  - Hematology & Oncology Associates of NEPA, Dunmore, Pennsylvania
  - Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - Hematology & Oncology Associates of NEPA, Scranton, Pennsylvania
  - Viewmont Medical Services, Scranton, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Mercy Health Partners, Scranton, Pennsylvania
  - Moses Taylor Hospital, Scranton, Pennsylvania
  - Associates in Hematology-Oncology, P.C., Upland, Pennsylvania
  - Roper Hospital-Department of Radiology, Charleston, South Carolina
  - Carolina Center of Gynecologic Oncology, PA, Charleston, South Carolina
  - South Carolina Oncology, Columbia, South Carolina
  - Greenville Hospital System, Greenville, South Carolina
  - Spartanburg Regional Healthcare System, Spartanburg, South Carolina
  - Sioux Valley Clinic - Clinical Research Center, Sioux Falls, South Dakota
  - Sioux Valley Clinic Oncology, Sioux Falls, South Dakota
  - Sioux Valley Hospital - North Center Radiology, Sioux Falls, South Dakota
  - Sioux Valley Clinic OBGYN, Ltd., Sioux Falls, South Dakota
  - The Family Cancer Center, Bartlett, Tennessee
  - Baroness Erlander Hospital, Chattanooga, Tennessee
  - Chattanooga GYN Oncology, Chattanooga, Tennessee
  - Parkridge Medical Center, Chattanooga, Tennessee
  - The Family Cancer Center, Collierville, Tennessee
  - The Family Cancer Center, Memphis, Tennessee
  - Arlington Cancer Center, Arlington, Texas
  - Center for Oncology Research and Treatment, PA, Dallas, Texas
  - Texas Cancer Associates, Dallas, Texas
  - Texas Cancer Associates, Plano, Texas
  - Center for Oncology Research and Treatment, PA, Richardson, Texas
  - Danville Hematology and Oncology, Inc., Danville, Virginia
  - VCU Health System at Stony Point, Richmond, Virginia
  - VCU Health System-Dalton Oncology Clinic, North Hospital, Richmond, Virginia
  - Carilion GYN Oncology Associates, Roanoke, Virginia
  - Western Washington Oncology, Inc., P.S., Aberdeen, Washington
  - Western Washington Oncology, Inc., P. S., Centralia, Washington
  - Covington MultiCare - Oncology Clinic, Covington, Washington
  - Gig Harbor Medical Oncology, Gig Harbor, Washington
  - Western Washington Oncology, Inc., P.S., Lacey, Washington
  - Western Washington Oncology, Inc., P.S., Shelton, Washington
  - Allenmore Hospital - Hematology Oncology Clinic, Tacoma, Washington
  - MultiCare Health System - Medical Oncology, Tacoma, Washington
  - Marshfield Clinic - Chippewa Falls Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Care - Regional Cancer Center - Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Marshfield Clinic - Lakeland Center, Minocqua, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - St. Michael's Hospital, Stevens Point, Wisconsin
  - Marchfield Clinic - Wausau Center, Wausau, Wisconsin
  - Marshfield Clinic Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin

REFERENCES:
- [Derived] Newhouse R, Nelissen E, El-Shakankery KH, Rogozinska E, Bain E, Veiga S, Morrison J. Pegylated liposomal doxorubicin for relapsed epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Jul 5;7(7):CD006910. doi: 10.1002/14651858.CD006910.pub3. PMID 37407274